CLINICAL TRIAL: NCT01758016
Title: Haptoglobin and Diabetes Complications in Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 2304-2000-RMB CTIL
Record Dates: First submitted 2012-12-23; First posted 2012-12-31 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes in Pregnancy
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Pregnancies of patients with Diabetes are associated with increase adverse pregnancy outcome . The risk for vascular complications including: Intra uterine growth restriction (20%), hypertension (31%), preeclampsia (15%), eclampsia and placental abruption are significantly greater than those in background populations. The risk of developing vascular complications in diabetes pregnancies although is correlated with the severity and length of the disease is not fully understood. Enhanced oxidation has been suggested to be the underlying abnormality responsible for some of the complications of diabetes.

Haptoglobin (Hp) is an abundant plasma glycoprotein produced in the liver. The best understood function of Hp is to bind free hemoglobin (Hb) released from red blood cells. Extracorpuscular Hb is a potent Fenton reagent.capable of of inflicting oxidative tissue damage. Hp binds to Hb and serves to inhibit the oxidative potential of Hb by preventing the release of heme iron.

The haptoglobin (Hp) gene at chromosomal locus 16q22 is polymorphic, with two common alleles denoted 1 and 2. the prevalence of Hp 1-1, Hp 1-2 and Hp 2-2 genotypes is approximately 16%, 48% and 36%, respectively. In the western world. A total of five independent longitudinal studies have demonstrated that DM individuals with Hp 2-2 genotype have a two to five-fold increased risk of CVD as compared to DM individuals without the Hp 2-2 genotype We sought to determine whether HP genotype plays important role in development of vascular complications in pregastational pregnancies. and whether Hp genotype 2-2 is a risk factor for developing gestational diabetes (GDM)

ELIGIBILITY:
Inclusion Criteria:

* Diabetes in pregnancy

Exclusion Criteria:

* Not willing to participate

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Pregastetional diabetic patients currently pregnant
  2. Gestational diabetes patients currently pregnant
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2012-11; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
vascular complications in pregnancy | 9 months

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Cmpus, Haifa
  - Meir Hospital, Kfar Saba